CLINICAL TRIAL: NCT02839330
Title: A Phase 3 Randomized, Observer-Blind, Multi-center, Controlled Study to Evaluate Safety, Immunogenicity, and Lot-to-Lot Consistency of an Adjuvanted Cell Culture-Derived, H5N1 Subunit Influenza Virus Vaccine in Healthy Adult Subjects ≥18 Years of Age
Brief Title: A Study to Evaluate Safety, Immunogenicity, and Lot-to-Lot Consistency of H5N1 Subunit Influenza Virus Vaccine in Healthy Adult Subjects ≥18 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V89_18
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Results first posted 2019-04-04 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2019-04

CONDITIONS: Avian Influenza
Keywords: Influenza; Vaccine; Flu; Avian; Pandemic; H5N1; MF59
MeSH Terms: conditions — Influenza in Birds; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): aH5N1c lot #1; receive 2 doses (on Day 1 and Day 22)
  Interventions: Biological: aH5N1c
- Group B (Experimental): aH5N1c lot #2; receive 2 doses (on Day 1 and Day 22)
  Interventions: Biological: aH5N1c
- Group C (Experimental): aH5N1c lot #3; receive 2 doses (on Day 1 and Day 22)
  Interventions: Biological: aH5N1c
- Group D (Placebo Comparator): Placebo; receive 2 doses (on Day 1 and Day 22)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: aH5N1c — Intramuscular (IM) administration, containing 7.5 mcg H5N1 hemagglutinin antigen (HA) + 0.25 mL MF59 (approximately 0.5 mL total volume).
  Arms: Group A; Group B; Group C
Biological: Placebo — Placebo: Saline injection
  Arms: Group D

SUMMARY:
This Phase 3 study evaluates the safety, immunogenicity and lot-to lot consistency of 3 lots of aH5N1c vaccine for pandemic avian influenza, in approximately 2394 healthy adults ≥18 years of age receiving the vaccine and 797 healthy adults receiving placebo. Subjects were randomized in a 3:1 ratio to receive either aH5N1c vaccine or saline placebo. Enrollment was stratified by age: 18 to <65 years of age and ≥65 years of age, to allow adequate safety assessment of the entire age spectrum.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years of age, mentally competent, in good health as determined by medical history, physical examination and clinical judgment by the Investigator; able to comply with all study procedures, to be contacted, and to be available for study visits according to the protocol.

Exclusion Criteria:

* Individuals who are pregnant or breastfeeding. Female subjects of childbearing potential must have a negative pregnancy test prior to study vaccines being administered.
* Females of childbearing potential who refuse to use an acceptable method of birth control from Day 1 (1st vaccination) to 3 weeks after the second study vaccination, and, if sexually active, who have not used a reliable birth control method for at least two months prior to study entry.
* Individuals with a body temperature ≥38.0 °C (≥100.4 °F) or any acute illness within 3 days of intended study vaccination.
* Individuals who received any type of influenza vaccine (e.g., "seasonal") within 7 days prior to enrolment in this study or who are planning to receive any type of influenza vaccine within 7 days (before or after) from the study vaccines.
* Individuals who received any other licensed vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this study or who are planning to receive any (non-influenza) vaccine within 28 days (before or after) from the study vaccines.
* Individuals with known or suspected impairment of the immune system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3196 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Director, Study Director — Seqirus
Locations (26):
- United States (26):
  - Optimal Research, LLC, Huntsville, Alabama
  - Radiant Research, Chandler, Arizona
  - Clinical Research Consortium Arizona, Tempe, Arizona
  - Optimal Research Site, San Diego, California
  - California Research Foundation, San Diego, California
  - Clinical Research Consulting, LLC, Milford, Connecticut
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Optimal Research, LLC, Melbourne, Florida
  - Great Lakes Clinical Trials LLC, Chicago, Illinois
  - Optimal Research, Peoria, Illinois
  - Heartland Research Associates, Wichita, Kansas
  - Optimal Research, LLC, Rockville, Maryland
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - RCR/United Medical Associates, PC, Binghamton, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - PMG Research of Raleigh, Raleigh, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Aventiv Research, Columbus, Ohio
  - Medical Research South, Charleston, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Biogenics Research Institute, San Antonio, Texas
  - J. Lewis Research Inc.-Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / FirstMed East, Salt Lake City, Utah
  - J. Lewis Research, Inc/Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Inc/Jordan River Family Medicine, South Jordan, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peterson J, Van Twuijver E, Versage E, Hohenboken M. Phase 3 Randomized, Multicenter, Placebo-Controlled Study to Evaluate Safety, Immunogenicity, and Lot-to-Lot Consistency of an Adjuvanted Cell Culture-Derived, H5N1 Subunit Influenza Virus Vaccine in Healthy Adult Subjects. Vaccines (Basel). 2022 Mar 23;10(4):497. doi: 10.3390/vaccines10040497. PMID 35455245

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 26 centers in the USA.
Pre-assignment Details: All enrolled subjects were included in the study. A total of 5 subjects were enrolled and randomized in error by sites. These subjects were deemed screen or randomization failures due to violation of the inclusion and/or exclusion criteria. Therefore, of the 3196 subjects enrolled in the study 3191 subjects were vaccinated.
Groups:
- Group A: aH5N1c Lot #1: aH5N1c lot #1; receive 2 doses (on Day 1 and Day 22)
- Group B: aH5N1c Lot #2: aH5N1c lot #2; receive 2 doses (on Day 1 and Day 22)
- Group C: aH5N1c Lot #3: aH5N1c lot #3; receive 2 doses (on Day 1 and Day 22)
- Group D: Placebo: Placebo; receive 2 doses (on Day 1 and Day 22)
Period: Overall Study
Arm/Group | Group A: aH5N1c Lot #1 | Group B: aH5N1c Lot #2 | Group C: aH5N1c Lot #3 | Group D: Placebo
Started (as randomized population) | 804 | 799 | 795 | 798
Exposed | 804 | 797 | 793 | 797
Completed | 746 | 741 | 747 | 747
Not Completed | 58 | 58 | 48 | 51
Not completed — Adverse Event | 0 | 1 | 2 | 2
Not completed — Death | 4 | 6 | 1 | 1
Not completed — Withdrawal by Subject | 27 | 19 | 11 | 13
Not completed — Lost to Follow-up | 22 | 27 | 29 | 25
Not completed — Administrative Reason | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 2 | 2 | 3
Not completed — Other reason, not specified | 4 | 3 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: aH5N1c Lot #1 | Group B: aH5N1c Lot #2 | Group C: aH5N1c Lot #3 | Group D: Placebo | Total
Number analyzed (Participants) | 804 | 799 | 795 | 798 | 3196
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 403 | 399 | 397 | 398 | 1597
  >=65 years | 401 | 400 | 398 | 400 | 1599
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (17.67) | 57.5 (17.83) | 57.5 (18.24) | 57.7 (18.29) | 57.7 (18.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 444 | 434 | 447 | 438 | 1763
  Male | 360 | 365 | 348 | 360 | 1433
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 53 | 61 | 64 | 55 | 233
  Not Hispanic or Latino | 746 | 729 | 721 | 732 | 2928
  Unknown or Not Reported | 5 | 9 | 10 | 11 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 4 | 5 | 3 | 18
  Asian | 12 | 7 | 9 | 7 | 35
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 1 | 4 | 10
  Black or African American | 110 | 102 | 104 | 112 | 428
  White | 668 | 679 | 674 | 665 | 2686
  More than one race | NA — Not assessed | NA — Not assessed | NA — Not assessed | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 5 | 5 | 2 | 7 | 19
Region of Enrollment [Number; unit: participants]
  United States | 804 | 799 | 795 | 798 | 3196
Weight [Mean (Standard Deviation); unit: kg] — Population: N=794 for aH5N1C lot#3 and 3195 for total for weight and height.
  kg
    number analyzed (Participants) | 804 | 799 | 794 | 798 | 3195
    (all) | 78.86 (15.049) | 80.22 (15.165) | 78.86 (15.302) | 79.84 (15.255) | 79.44 (15.197)
Height [Mean (Standard Deviation); unit: cm] — Population: N=794 for aH5N1C lot#3 and 3195 for total for weight and height.
  cm
    number analyzed (Participants) | 804 | 799 | 794 | 798 | 3195
    (all) | 169.38 (9.596) | 169.37 (9.708) | 169.37 (10.153) | 169.78 (9.424) | 169.47 (9.720)

OUTCOME MEASURES:

1. Primary Outcome: Primary Immunogenicity Endpoint: Geometric Mean Titer (GMT) at Day 43 by Lot
Description: Hemagglutination Inhibition (HI) GMT was assessed at Day 1 and Day 43 for 3 consecutively produced lots.
Time Frame: Day 1, Day 43
Population: Per Protocol Set (PPS) - All subjects who received at least one dose of study vaccination and provided at least one evaluable serum sample (lot-to-lot consistency) at relevant timepoints and who correctly received the vaccine, had no major protocol deviations leading to exclusion, and were not excluded due to other reasons.
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | Group A: aH5N1c Lot #1 | Group B: aH5N1c Lot #2 | Group C: aH5N1c Lot #3
Number analyzed (Participants) | 761 | 747 | 741
geometric mean titer
  Day 1 | 16.1 [15.1 to 17.2] | 17.0 [15.9 to 18.2] | 17.0 [15.9 to 18.2]
  Day 43: number analyzed (Participants) | 729 | 710 | 717
  Day 43 | 128.6 [118.9 to 139.1] | 127.4 [117.6 to 138.0] | 132.2 [122.1 to 143.1]
Statistical Analysis 1: Comparison: Group A: aH5N1c Lot #1 vs Group B: aH5N1c Lot #2; aH5N1c Lot #1 vs. aH5N1c Lot #2; Test type: Equivalence — Equivalence margin: The 2-sided 95% confidence interval (CI) of all the 3 pairwise comparisons of GMTs to fall between the predefined equivalence ranges of 0.667 and 1.5; GMT ratio = 1.01, 95% CI 2-sided [0.90 to 1.13]
Statistical Analysis 2: Comparison: Group B: aH5N1c Lot #2 vs Group C: aH5N1c Lot #3; aH5N1c Lot #2 vs. aH5N1c Lot #3; Test type: Equivalence — Equivalence margin: The 2-sided 95% CIs of all the 3 pairwise comparisons of GMTs to fall between the predefined equivalence ranges of 0.667 and 1.5; GMT ratio = 0.96, 95% CI 2-sided [0.86 to 1.08]
Statistical Analysis 3: Comparison: Group A: aH5N1c Lot #1 vs Group C: aH5N1c Lot #3; aH5N1c Lot #1 vs. aH5N1c Lot #3; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; GMT ratio = 0.97, 95% CI 2-sided [0.87 to 1.09]

2. Primary Outcome: Primary Immunogenicity Endpoint: Percentage of Subjects With Haemagglutination Inhibition (HI) Titer ≥ 1:40 at Day 43 by Age Cohort
Description: Percentage of subjects with HI titer ≥ 1:40 at Day 43 was assessed by age cohort (18 to <65 years of age and ≥65 years of age) for the pooled lots. Center for Biologics Evaluation and Research (CBER) criterion for subjects aged 18 to <65 years: The lower bound of the 2-sided 95% CI for the percentage of subjects achieving an HI antibody titer ≥1:40 should meet or exceed 70%. CBER criterion for subjects aged ≥65 years: The lower bound of the 2-sided 95% CI for the percentage of subjects achieving an HI antibody titer ≥1:40 should meet or exceed 60%.
Time Frame: Day 1, Day 43
Population: The PPS consisting of all subjects who received at least one dose of study vaccination and provided at least one evaluable serum sample at relevant timepoints who correctly received the vaccine, had no major protocol deviations leading to exclusion, and were not excluded due to other reasons was used for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- aH5N1c: aH5N1c (Active Treatment Groups); receive 2 doses (on Day 1 and Day 22)
- Placebo: Placebo; receive 2 doses (on Day 1 and Day 22)
Arm/Group | aH5N1c | Placebo
Number analyzed (Participants) | 2249 | 739
percentage of subjects
  Day 1, 18 to <65 years: number analyzed (Participants) | 1116 | 372
  Day 1, 18 to <65 years | 13.0 [10.7 to 15.6] | 15.0 [11.5 to 19.4]
  Day 1, ≥65 Years: number analyzed (Participants) | 1133 | 367
  Day 1, ≥65 Years | 27.8 [24.9 to 30.9] | 24.5 [20.1 to 29.6]
  Day 43, 18 to <65 years: number analyzed (Participants) | 1076 | 349
  Day 43, 18 to <65 years | 95.0 [93.4 to 96.2] | 8.5 [5.9 to 12.1]
  Day 43, ≥65 Years: number analyzed (Participants) | 1080 | 351
  Day 43, ≥65 Years | 85.7 [83.3 to 87.9] | 20.8 [16.6 to 25.8]

3. Primary Outcome: Percentage of Subjects With Solicited Local, Solicited Systemic, and Other Adverse Events (AEs) as Measured for 7 Days (Inclusive) Following Each Vaccination
Description: Percentages of subjects with solicited local, solicited systemic, and other AEs as measured for 7 days (inclusive) following each vaccination (first and second) and any (first or second) vaccination, by treatment group and calculated for several time intervals after vaccination : 30 minutes, 1 to 3 days (without 30 minutes), 4 to 7 days, and 1 to 7 days (without 30 minutes), and 1 to 3 days (including 30 minutes) and 1 to 7 days (including 30 minutes). Analysis for intervals of the first 30 minutes, days 1 to 3, and days 4 to 7 was not performed.
Time Frame: Day 1 to Day 7
Population: The overall safety set consisting of all subjects who received a study vaccination who underwent any assessment of local and systemic site reaction and/or assessment of any use of analgesics/antipyretics was used for analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | aH5N1c | Placebo
Number analyzed (Participants) | 2395 | 796
percentage of subjects
  Any Solicited AE, After Any Vac (D1-D7 excl 30m): number analyzed (Participants) | 2352 | 784
  Any Solicited AE, After Any Vac (D1-D7 excl 30m) | 59.7 | 38.0
  Solicited Loc AE, After Any Vac (D1-D7 excl 30m): number analyzed (Participants) | 2352 | 784
  Solicited Loc AE, After Any Vac (D1-D7 excl 30m) | 50.2 | 14.7
  Solicited Sys AE, After Any Vac (D1-D7 excl 30m): number analyzed (Participants) | 2352 | 784
  Solicited Sys AE, After Any Vac (D1-D7 excl 30m) | 38.2 | 32.8
  Any Solicited AE, After Vac 1 (D1-D7 excl 30m): number analyzed (Participants) | 2346 | 782
  Any Solicited AE, After Vac 1 (D1-D7 excl 30m) | 52.4 | 30.2
  Solicited Loc AE, After Vac 1 (D1-D7 excl 30m): number analyzed (Participants) | 2346 | 782
  Solicited Loc AE, After Vac 1 (D1-D7 excl 30m) | 43.2 | 10.2
  Solicited Sys AE, After Vac 1 (D1-D7 excl 30m): number analyzed (Participants) | 2346 | 770
  Solicited Sys AE, After Vac 1 (D1-D7 excl 30m) | 30.7 | 26.0
  Any Solicited AE, After Vac 2 (D1-D7 excl 30m): number analyzed (Participants) | 2304 | 770
  Any Solicited AE, After Vac 2 (D1-D7 excl 30m) | 41.1 | 22.3
  Solicited Loc AE, After Vac 2 (D1-D7 excl 30m): number analyzed (Participants) | 2304 | 770
  Solicited Loc AE, After Vac 2 (D1-D7 excl 30m) | 33.9 | 7.4
  Solicited Sys AE, After Vac 2 (D1-D7 excl 30m): number analyzed (Participants) | 2304 | 770
  Solicited Sys AE, After Vac 2 (D1-D7 excl 30m) | 21.3 | 18.6
  Any Solicited AE, After Any Vac (D1-D7) | 59.3 | 38.7
  Solicited Loc AE, After Any Vac (D1-D7) | 50.0 | 16.3
  Solicited Sys AE, After Any Vac (D1-D7) | 37.7 | 32.5
  Any Solicited AE, After Vac 1 (D1-D7) | 52.0 | 30.3
  Solicited Loc AE, After Vac 1 (D1-D7) | 42.8 | 11.1
  Solicited Sys AE, After Vac 1 (D1-D7) | 30.3 | 25.5
  Any Solicited AE, After Vac 2 (D1-D7): number analyzed (Participants) | 2334 | 779
  Any Solicited AE, After Vac 2 (D1-D7) | 41.0 | 23.1
  Solicited Loc AE, After Vac 2 (D1-D7): number analyzed (Participants) | 2334 | 779
  Solicited Loc AE, After Vac 2 (D1-D7) | 34.1 | 8.3
  Solicited Sys AE, After Vac 2 (D1-D7): number analyzed (Participants) | 2334 | 779
  Solicited Sys AE, After Vac 2 (D1-D7) | 21.2 | 18.9

4. Primary Outcome: Percentages of Subjects With Any Unsolicited AEs Reported Through 21 Day After Vaccination
Description: Percentages of subjects with any unsolicited AEs reported through 21 days after each (first and second) and any (first or second) vaccination by treatment group.
Time Frame: Day 1 to Day 43
Population: The unsolicited safety set consisting of all subjects who received a study vaccination and who underwent any AEs assessment (ie, a subject did not have to have any AEs) was used for analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | aH5N1c | Placebo
Number analyzed (Participants) | 2395 | 796
percentage of subjects
  Unsolicited AEs, V1 or V2 | 23.4 | 22.2
  Possibly/probably related unsolicited AE, V1 or V2 | 7.0 | 6.2
  Unsolicited AE, V1 | 15.3 | 13.2
  Possibly/probably related unsolicited AE, V1 | 4.8 | 3.8
  Unsolicited AE, V2 | 12.2 | 11.9
  Possibly/probably related unsolicited AE, V2 | 2.8 | 2.8

5. Primary Outcome: Percentages of Subjects Reporting SAEs, AESIs, NOCD, AEs Leading to Vaccine/Study Withdrawal, and Medically Attended AEs, and Concomitant Medications Associated With These Events as Collected From Day 1 to Day 387, by Vaccine Group.
Description: Percentages of subjects with any adverse events (AE), adverse events of special interest (AESI), new onset of chronic disease (NOCD), and serious adverse event (SAE) through study termination by treatment group.
Time Frame: Day 1 to Day 387
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | aH5N1c | Placebo
Number analyzed (Participants) | 2395 | 796
percentage of subjects
  SAE | 6.7 | 9.3
  Possibly or probably related SAEs | 0 | 0.3
  AEs leading to premature withdrawal | 0.5 | 0.4
  Medically attended AEs | 46.5 | 46.0
  AEs leading to NOCD | 9.5 | 9.2
  AESI | 0.3 | 0.9
  AE leading to death | 0.5 | 0.1

6. Secondary Outcome: Secondary Immunogenicity Endpoint: Geometric Mean Titer (GMT) at Day 1, Day 22, Day 43, and Day 183 by Vaccine Group (aH5N1c or Placebo) and by Age Cohort (18 to <65 Years of Age and ≥65 Years of Age).
Description: Estimates of hemagglutination inhibition (HI) GMTs, and their associated 95% CIs at Day 1, Day 22, Day 43 and Day 183 were computed using ANCOVA with factors for treatment (active treatment groups or placebo), center and a covariate for the effect defined by the log-transformed prevaccination antibody titer (Day 1).
Time Frame: Day 1, Day 22, Day 43, and Day 183
Population: PPS - All subjects who received at least one dose of study vaccination and provided at least one evaluable serum sample at relevant timepoints and who correctly received the vaccine, had no major protocol deviations leading to exclusion, and were not excluded due to other reasons.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- aH5N1c: aH5N1c: Active Treatment Groups, received 2 doses on Day 1 and Day 22
- Placebo: Placebo, received 2 doses on Day 1 and Day 22
Arm/Group | aH5N1c | Placebo
Number analyzed (Participants) | 2249 | 739
titer
  Day 1 | 16.6 [16.0 to 17.3] | 16.7 [15.6 to 17.9]
  Day 1, 18 to <65 years: number analyzed (Participants) | 1116 | 372
  Day 1, 18 to <65 years | 13.5 [12.8 to 14.2] | 13.7 [12.5 to 15.0]
  Day 1, ≥65 years: number analyzed (Participants) | 1133 | 367
  Day 1, ≥65 years | 20.5 [19.4 to 21.8] | 20.6 [18.6 to 22.7]
  Day 22: number analyzed (Participants) | 2245 | 736
  Day 22 | 46.4 [44.5 to 48.4] | 13.0 [12.1 to 14.0]
  Day 22, 18 to <65 years: number analyzed (Participants) | 1115 | 370
  Day 22, 18 to <65 years | 50.6 [47.6 to 53.8] | 11.6 [10.4 to 12.9]
  Day 22, ≥65 years: number analyzed (Participants) | 1130 | 366
  Day 22, ≥65 years | 42.4 [40.0 to 45.0] | 14.5 [13.1 to 16.0]
  Day 43: number analyzed (Participants) | 2156 | 700
  Day 43 | 130.6 [124.8 to 136.6] | 13.7 [12.6 to 14.8]
  Day 43, 18 to <65 years: number analyzed (Participants) | 1076 | 349
  Day 43, 18 to <65 years | 170.7 [160.5 to 181.6] | 11.0 [9.9 to 12.2]
  Day 43, ≥65 years: number analyzed (Participants) | 1080 | 351
  Day 43, ≥65 years | 97.9 [92.1 to 104.1] | 16.7 [15.0 to 18.5]
  Day 183: number analyzed (Participants) | 2079 | 687
  Day 183 | 20.0 [19.2 to 20.8] | 7.7 [7.2 to 8.2]
  Day 183, 18 to <65 years: number analyzed (Participants) | 1025 | 341
  Day 183, 18 to <65 years | 20.4 [19.3 to 21.6] | 6.8 [6.1 to 7.4]
  Day 183, ≥65 years: number analyzed (Participants) | 1054 | 346
  Day 183, ≥65 years | 19.3 [18.2 to 20.4] | 8.6 [7.8 to 9.5]

7. Secondary Outcome: Secondary Immunogenicity Endpoint: Percentage of Subjects With Haemagglutination Inhibition (HI) Titer ≥ 1:40 on Day 1, Day 22, Day 43 and Day 183 by Vaccine Group (aH5N1c or Placebo) and by Age Cohort (18 to <65 Years of Age and ≥65 Years of Age).
Description: The percentage of subjects with HI titer ≥1:40 data over time by vaccine group and age cohort are presented. CBER criterion for subjects aged 18 to <65 years: The lower bound of the 2-sided 95% CI for the percentage of subjects achieving an HI antibody titer ≥1:40 should meet or exceed 70%.
  CBER criterion for subjects aged ≥65 years: The lower bound of the 2-sided 95% CI for the percentage of subjects achieving an HI antibody titer ≥1:40 should meet or exceed 60%.
Time Frame: Day 1, Day 22, Day 43 and Day 183
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | aH5N1c | Placebo
Number analyzed (Participants) | 2249 | 739
percentage of subjects
  Day 1 | 22.9 [21.1 to 24.6] | 22.6 [19.6 to 25.8]
  Day 1, 18 to <65 years: number analyzed (Participants) | 1116 | 372
  Day 1, 18 to <65 years | 17.4 [15.2 to 19.7] | 19.6 [15.7 to 24.0]
  Day 1, ≥65 years: number analyzed (Participants) | 1133 | 367
  Day 1, ≥65 years | 28.2 [25.6 to 31.0] | 25.6 [21.2 to 30.4]
  Day 22: number analyzed (Participants) | 2245 | 736
  Day 22 | 59.3 [57.2 to 61.3] | 14.9 [12.4 to 17.7]
  Day 22, 18 to <65 years: number analyzed (Participants) | 1115 | 370
  Day 22, 18 to <65 years | 63.0 [60.1 to 65.9] | 13.5 [10.2 to 17.4]
  Day 22, ≥65 years: number analyzed (Participants) | 1130 | 366
  Day 22, ≥65 years | 55.6 [52.6 to 58.5] | 16.4 [12.7 to 20.6]
  Day 43: number analyzed (Participants) | 2156 | 700
  Day 43 | 88.3 [86.9 to 89.6] | 16.9 [14.2 to 19.8]
  Day 43, 18 to <65 years: number analyzed (Participants) | 1076 | 349
  Day 43, 18 to <65 years | 93.1 [91.4 to 94.6] | 10.9 [7.8 to 14.6]
  Day 43, ≥65 years: number analyzed (Participants) | 1080 | 351
  Day 43, ≥65 years | 83.5 [81.2 to 85.7] | 22.8 [18.5 to 27.5]
  Day 183: number analyzed (Participants) | 2079 | 687
  Day 183 | 32.6 [30.6 to 34.6] | 5.2 [3.7 to 7.2]
  Day 183, 18 to <65 years: number analyzed (Participants) | 1025 | 341
  Day 183, 18 to <65 years | 34.2 [31.3 to 37.2] | 2.1 [0.8 to 4.2]
  Day 183, ≥65 years: number analyzed (Participants) | 1054 | 346
  Day 183, ≥65 years | 30.9 [28.1 to 33.8] | 8.4 [5.7 to 11.8]

8. Secondary Outcome: Secondary Immunogenicity Endpoint: Percentage of Subjects Achieving Seroconversion on Day 22, and Day 43 by Vaccine Group (aH5N1c or Placebo) and by Age Cohort (18 to <65 Years of Age and ≥65 Years of Age).
Description: Percentage of subjects achieving seroconversion (defined as: HI titer ≥1:40 for subjects negative at baseline [HI titer <1:10]; or a minimum 4-fold increase in HI titer for subjects positive at baseline [HI titer ≥1:10]) on Day 22, and Day 43 by vaccine group (aH5N1c or placebo) and by age cohort (18 to <65 years of age and ≥65 years of age).
Time Frame: Day 22, and Day 43
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | aH5N1c | Placebo
Number analyzed (Participants) | 2249 | 739
percentage of subjects
  Day 22: number analyzed (Participants) | 2245 | 736
  Day 22 | 32.2 [30.3 to 34.2] | 1.1 [0.5 to 2.1]
  Day 22, 18 to <65 years: number analyzed (Participants) | 1115 | 370
  Day 22, 18 to <65 years | 40.4 [37.6 to 43.4] | 1.9 [0.8 to 3.9]
  Day 22, ≥65 years: number analyzed (Participants) | 1130 | 366
  Day 22, ≥65 years | 24.2 [21.7 to 26.8] | 0.3 [0.0 to 1.5]
  Day 43: number analyzed (Participants) | 2156 | 700
  Day 43 | 66.9 [64.9 to 68.9] | 1.0 [0.4 to 2.0]
  Day 43, 18 to <65 years: number analyzed (Participants) | 1076 | 349
  Day 43, 18 to <65 years | 79.9 [77.4 to 82.3] | 0.3 [0.0 to 1.6]
  Day 43, ≥65 Years: number analyzed (Participants) | 1080 | 351
  Day 43, ≥65 Years | 54.0 [51.0 to 57.0] | 1.7 [0.6 to 3.7]

9. Secondary Outcome: Secondary Immunogenicity Endpoint: Geometric Mean Titer (GMT) at Day 1, Day 22, Day 43 and Day 183 by Vaccine Group (aH5N1c or Placebo) and By Age Cohort (18 to <60 Years of Age and ≥60 Years of Age)
Description: Hemagglutination inhibition (HI) GMTs were assessed over time for the vaccine group and age cohort. Adjusted estimates of GMTs, and their associated 95% CIs at Day 1, Day 22, Day 43 and Day 183 were computed using ANCOVA with factors for treatment (active treatment groups or placebo), center and a covariate for the effect defined by the log-transformed prevaccination antibody titer (Day 1).
Time Frame: Day 1, Day 22, Day 43 and Day 183
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: titer
Arm/Group | aH5N1c | Placebo
Number analyzed (Participants) | 2249 | 739
titer
  Day 1, 18 to <60 years: number analyzed (Participants) | 980 | 331
  Day 1, 18 to <60 years | 13.0 [12.3 to 13.8] | 13.4 [12.2 to 14.7]
  Day 1, ≥60 years: number analyzed (Participants) | 1269 | 408
  Day 1, ≥60 years | 20.1 [19.1 to 21.3] | 20.1 [18.3 to 22.0]
  Day 22, 18 to <60 years: number analyzed (Participants) | 979 | 329
  Day 22, 18 to <60 years | 51.1 [47.9 to 54.6] | 11.2 [10.0 to 12.5]
  Day 22, ≥60 years: number analyzed (Participants) | 1266 | 407
  Day 22, ≥60 years | 42.9 [40.5 to 45.3] | 14.4 [13.1 to 15.9]
  Day 43, 18 to <60 years: number analyzed (Participants) | 947 | 309
  Day 43, 18 to <60 years | 177.4 [166.2 to 189.4] | 10.7 [9.5 to 11.9]
  Day 43, ≥60 years: number analyzed (Participants) | 1209 | 391
  Day 43, ≥60 years | 100.7 [95.0 to 106.7] | 16.2 [14.7 to 17.9]
  Day 183, 18 to <60 years: number analyzed (Participants) | 899 | 302
  Day 183, 18 to <60 years | 20.4 [19.3 to 21.7] | 6.7 [6.0 to 7.4]
  Day 183, ≥60 years: number analyzed (Participants) | 1180 | 385
  Day 183, ≥60 years | 19.3 [18.3 to 20.4] | 8.5 [7.7 to 9.3]

10. Secondary Outcome: Secondary Immunogenicity Endpoint: Percentage of Subjects With Haemagglutination Inhibition (HI) Titer ≥ 1:40 on Day 1, Day 22, Day 43, and Day 183 by Vaccine Group (aH5N1c or Placebo) and by Age Cohort (18 to <60 Years of Age and ≥60 Years of Age)
Description: The percentage of subjects with HI titer ≥1:40 data over time by vaccine group and age cohort. Committee for Medicinal Products for Human Use (CHMP) criterion for subjects aged 18 to <60 years: The percentage of subjects achieving an HI titer ≥1:40 is >70%. CHMP criterion for subjects aged ≥60 years: The percentage of subjects achieving an HI titer ≥1:40 is >60%.
Time Frame: Day 1, Day 22, Day 43, and Day 183
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | aH5N1c | Placebo
Number analyzed (Participants) | 2249 | 739
percentage of subjects
  Day 1, 18 to <60 years: number analyzed (Participants) | 980 | 331
  Day 1, 18 to <60 years | 17.1 [14.8 to 19.7] | 19.6 [15.5 to 24.3]
  Day 1, ≥60 years: number analyzed (Participants) | 1269 | 408
  Day 1, ≥60 years | 27.3 [24.8 to 29.8] | 25.0 [20.9 to 29.5]
  Day 22, 18 to <60 years: number analyzed (Participants) | 979 | 329
  Day 22, 18 to <60 years | 63.2 [60.1 to 66.3] | 12.2 [8.8 to 16.2]
  Day 22, ≥60 years: number analyzed (Participants) | 1266 | 407
  Day 22, ≥60 years | 56.2 [53.5 to 59.0] | 17.2 [13.7 to 21.2]
  Day 43, 18 to <60 years: number analyzed (Participants) | 947 | 309
  Day 43, 18 to <60 years | 93.6 [91.8 to 95.0] | 10.0 [6.9 to 13.9]
  Day 43, ≥60 years: number analyzed (Participants) | 1209 | 391
  Day 43, ≥60 years | 84.2 [82.0 to 86.2] | 22.3 [18.2 to 26.7]
  Day 183, 18 to <60 years: number analyzed (Participants) | 899 | 302
  Day 183, 18 to <60 years | 34.3 [31.2 to 37.5] | 2.3 [0.9 to 4.7]
  Day 183, ≥60 years: number analyzed (Participants) | 1180 | 385
  Day 183, ≥60 years | 31.3 [28.6 to 34.0] | 7.5 [5.1 to 10.6]

11. Secondary Outcome: Secondary Immunogenicity Endpoint: Percentage of Subjects Achieving Seroconversion on Day 22, and Day 43 by Vaccine Group (aH5N1c or Placebo) and by Age Cohort (18 to <60 Years of Age and ≥60 Years of Age)
Description: Percentage of subjects achieving seroconversion (defined as: HI titer ≥1:40 for subjects negative at baseline [HI titer <1:10]; or a minimum 4-fold increase in HI titer for subjects positive at baseline [HI titer ≥1:10]) on Day 22, and Day 43 by vaccine group (aH5N1c or placebo) and by age cohort (18 to <60 years of age and ≥60 years of age)
Time Frame: Day 22, and Day 43
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | aH5N1c | Placebo
Number analyzed (Participants) | 2249 | 739
percentage of subjects
  Day 22, 18 to <60 years: number analyzed (Participants) | 979 | 329
  Day 22, 18 to <60 years | 42.2 [39.1 to 45.4] | 1.5 [0.5 to 3.5]
  Day 22, ≥60 years: number analyzed (Participants) | 1266 | 407
  Day 22, ≥60 years | 24.6 [22.2 to 27.0] | 0.7 [0.2 to 2.1]
  Day 43, 18 to <60 years: number analyzed (Participants) | 947 | 309
  Day 43, 18 to <60 years | 81.6 [79.0 to 84.0] | 0.3 [0.0 to 1.8]
  Day 43, ≥60 years: number analyzed (Participants) | 1209 | 391
  Day 43, ≥60 years | 55.4 [52.6 to 58.2] | 1.5 [0.6 to 3.3]

12. Secondary Outcome: Secondary Immunogenicity Endpoint: Geometric Mean Ratio (GMR) of Haemagglutination Inhibition (HI) Titer: Day 22/Day 1, Day 43/Day 1 by Vaccine Group (aH5N1c or Placebo) and by Age Cohort (18 to <60 Years of Age and ≥60 Years of Age)
Description: The GMR of HI titers (Day 22/Day 1, Day 43/Day 1) is presented for the vaccine groups and age cohort. CHMP criterion for subjects aged 18 to <60 years: GMR is >2.5. CHMP criterion for subjects aged ≥60 years: GMR is >2.0.
Time Frame: Day 1, Day 22, Day 43
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | aH5N1c | Placebo
Number analyzed (Participants) | 2249 | 739
ratio
  Day 22/Day 1, Overall: number analyzed (Participants) | 2245 | 736
  Day 22/Day 1, Overall | 2.86 [2.74 to 2.98] | 0.80 [0.77 to 0.90]
  Day 43/Day 1, Overall: number analyzed (Participants) | 2156 | 700
  Day 43/Day 1, Overall | 7.96 [7.61 to 8.33] | 0.83 [0.74 to 0.86]
  Day 22/Day 1, 18 to <60 years: number analyzed (Participants) | 979 | 329
  Day 22/Day 1, 18 to <60 years | 3.92 [3.67 to 4.18] | 0.85 [0.76 to 0.96]
  Day 22/Day 1, ≥60 years: number analyzed (Participants) | 1266 | 407
  Day 22/Day 1, ≥60 years | 2.22 [2.10 to 2.35] | 0.75 [0.68 to 0.82]
  Day 43/Day 1, 18 to <60 years: number analyzed (Participants) | 947 | 309
  Day 43/Day 1, 18 to <60 years | 13.44 [12.59 to 14.35] | 0.81 [0.72 to 0.90]
  Day 43/Day 1, ≥60 years: number analyzed (Participants) | 1209 | 391
  Day 43/Day 1, ≥60 years | 5.18 [4.88 to 5.49] | 0.83 [0.76 to 0.92]

ADVERSE EVENTS:
Time Frame: Day 1 to Day 387
Description: The unsolicited safety set consisting of all subjects who received a study vaccination with documented safety assessments for unsolicited AE data (including those where it was reported/confirmed that no events had occurred).
  After lot-to-lot consistency was demonstrated, the populations of all aH5N1c vaccine recipients were pooled in order to evaluate immunogenicity and safety. Therefore, the H5N1c arms are pooled for the safety assessments.
Arm/Group | aH5N1c | Placebo
All-Cause Mortality (participants affected / at risk) | 11/2395 | 1/796
Serious Adverse Events (participants affected / at risk) | 161/2395 | 74/796
Other Adverse Events (participants affected / at risk) | 91/2395 | 44/796
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | aH5N1c (N=2395) | Placebo (N=796)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 8 | 8
Coronary artery disease (Cardiac disorders) | 3 | 3
Myocardial infarction (Cardiac disorders) | 2 | 4
Acute myocardial infarction (Cardiac disorders) | 4 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 3
Angina pectoris (Cardiac disorders) | 3 | 0
Atrial flutter (Cardiac disorders) | 2 | 0
Atrioventricular block (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Hypertensive heart disease (Cardiac disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac perforation (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 1
Gastritis alcoholic (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0
Coeliac disease (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Perforated ulcer (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Biliary cirrhosis primary (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0
Food allergy (Immune system disorders) | 1 | 0
Sarcoidosis (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 2
Diverticulitis (Infections and infestations) | 2 | 1
Appendicitis (Hepatobiliary disorders) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
External ear cellulitis (Infections and infestations) | 1 | 0
Gallbladder abscess (Infections and infestations) | 1 | 0
Incision site cellulitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Metapneumovirus infection (Infections and infestations) | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Shigella infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 4 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 0
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 15 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 2 | 3
Transient ischaemic attack (Nervous system disorders) | 3 | 1
Carotid artery stenosis (Nervous system disorders) | 2 | 1
Basal ganglia infarction (Nervous system disorders) | 1 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Cerebellar stroke (Nervous system disorders) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Acute psychosis (Psychiatric disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1
Borderline personality disorder (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Adenomyosis (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Hospitalisation (Surgical and medical procedures) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 2
Aortic aneurysm (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | aH5N1c (N=2395) | Placebo (N=796)
Upper respiratory tract infection (Infections and infestations) | 91 | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT02839330/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT02839330/SAP_001.pdf